CLINICAL TRIAL: NCT07171593
Title: Efficacy of High-protein Oral Enteral Nutrition Supplement Supplemented With HMB in Active Crohn's Disease With Sarcopenia: a Prospective, Randomized, Controlled Study
Brief Title: High-protein Oral Nutrition With HMB for Active CD Patients With Sarcopenia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chao Kang, Clinical professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-077
Record Dates: First submitted 2025-04-10; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Handgrip Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): EEN
- Experiment (Experimental): EEN+HMB
  Interventions: Dietary Supplement: HMB

INTERVENTIONS:
Dietary Supplement: HMB — EEN+HMB
  Arms: Experiment

SUMMARY:
The efficacy of B-hydroxy-β-methybutyrate in sarcopenia

ELIGIBILITY:
Inclusion Criteria:

1. Patients with active Crohn's disease (CD) who visited the Sixth Affiliated Hospital of Sun Yat-sen University between July 2023 and December 2024;
2. Aged 18-50 years;
3. Complicated with sarcopenia;
4. Willing and able to tolerate oral exclusive enteral nutrition (EEN) therapy;
5. Signed informed consent and able to comply with the study procedures;
6. Colonic or ileocolonic type CD (SES-CD ≥6; if only terminal ileum is involved, SES-CD ≥4).

Exclusion Criteria:

1. Short bowel syndrome;
2. High-output jejunal fistula;
3. Severe stress or shock status;
4. Complete mechanical intestinal obstruction, acute gastrointestinal bleeding, or severe intra-abdominal infection;
5. Severe hepatic, renal, or cardiac diseases, or malignant tumors;
6. History of allergy or contraindication to Ensure or HMB;
7. Persistent severe vomiting or intractable diarrhea;
8. Congenital disorders of sugar or amino acid metabolism;
9. Underwent CD-related intestinal surgery or received biologic therapy within the past month, or received immunosuppressive/antibiotic therapy related to CD within 2 weeks prior to enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
muscle strength improvement | Week 4; Week 8
  Grip strength was measured using an electronic dynamometer. Participants sat in an armchair with the upper arm in the adducted neutral position, the elbow flexed at 90°, and the forearm and wrist relaxed naturally. The test hand held the dynamometer and was instructed to squeeze with maximal force smoothly until reaching the peak value, without any twisting or jerking movements of the forearm or hand. After completing the measurement, the other hand was tested using the same method. Each trial was performed three times per hand with a one-minute interval between trials. The maximum value among the six trials was recorded as the final result.

SECONDARY OUTCOMES:
Improvement of muscle mass | Week 4; Week 8
  Appendicular skeletal muscle mass (ASM) was assessed in this study using a body composition analyzer. ASM was defined as the sum of muscle mass in the arms and legs. During the measurement, patients were required to fast, empty their bowels and bladder, wear light clothing, and undergo the test before exercise, bathing, or showering. Female patients were instructed to avoid measurements during menstruation.
Clinical response | Week 4; Week 8
  A decrease in the Crohn's Disease Activity Index (CDAI) by ≥70 points or a CDAI <150.
Clinical remission | Week 4; Week 8
  CDAI <150.
Mucosal healing | Week 4; Week 8
  No visible ulcers on endoscopy.
Clinical relapse | Week 4; Week 8
  CDAI ≥250 at any visit, or CDAI between 150-250 at two consecutive visits one week apart, with an increase of at least 70 points, accompanied by either CRP >5 mg/L or fecal calprotectin >250 μg/g.

CONTACTS AND LOCATIONS:
Overall Officials: Kang Chao, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Hospital Affiliated to Sun Yat-sen University, Guangzhou, Guangdong, China